CLINICAL TRIAL: NCT00319046
Title: Open-label, Non Comparative, Multi-center Study to Evaluate the Long Term Efficacy, Safety and Tolerability of Oral Miglustat as a Maintenance Therapy After a Switch From Enzyme Replacement Therapy in Adult Patients With Stable Type 1 Gaucher Disease
Brief Title: Clinical Study to Evaluate the Long Term Efficacy, Safety and Tolerability of Miglustat in Patients With Stable Type 1 Gaucher Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OGT 918-011
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Results first posted 2012-05-23 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Gaucher Disease Type 1
Keywords: enzyme replacement therapy; Type 1 Gaucher Disease; miglustat
MeSH Terms: conditions — Gaucher Disease | interventions — miglustat

ARMS (1):
- Open-label miglustat (Experimental): Oral administration of miglustat 100 mg t.i.d. for a period of 2 years
  Interventions: Drug: Miglustat

INTERVENTIONS:
Drug: Miglustat — Oral capsules containing miglustat 100 mg, administered three times daily (t.i.d.)
  Other Names: Zavesca

SUMMARY:
Although miglustat has been approved as a treatment for mild to moderate type 1 Gaucher disease in patients who are unsuitable for enzyme replacement therapy (ERT), more data are required to establish the long term efficacy, safety and tolerability of miglustat in maintaining diseases stability after a switch from ERT.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18 years or older
2. Type 1 Gaucher disease, diagnosed by glucocerebrosidase assay or molecular analysis of the glucocerebrosidase gene.
3. Treatment with ERT for at least 3 years, with a stable dose regimen for at least the last 6 months.
4. Clinically and biologically stable disease for the previous 2 years, with at least 2 time points assessments (including baseline as one potential time point), defined as:

   * Stable organomegaly (assessed by magnetic resonance imaging (MRI) or computed tomography (CT)):

     * Liver volume within 10% of the mean.
     * Spleen volume within 10% of the mean.
   * Free of progressive symptomatic documented bone disease.
   * Hemoglobin levels > 11g/dl
   * Mean platelet count > 100x10^9 /l.
   * Chitotriosidase activity within 20% of the mean.

     * If chitotriosidase is not available (in the case of chitotriosidase deficiency, or if it was not determined), other relevant biomarkers (e.g., angiotensin converting enzyme (ACE), tartrate resistant acid phosphatase (TRAP) and ferritin) could be considered.
5. Written informed consent.

Exclusion Criteria:

1. History or evidence of oculomotor gaze palsy, ataxia or other clinical manifestations typically associated with neuronopathic type 3 Gaucher disease.
2. Not ambulant patients, or with progressive symptomatic documented bone disease.
3. Splenectomy before 18 years of age for splenomegaly and/or thrombocytopenia.
4. Peripheral polyneuropathy (not mononeuropathy) documented with both clinical signs and symptoms, and electrodiagnostic (EDX).
5. Patients (males and females) who do not agree to use reliable contraception throughout the study and for 3 months after cessation of miglustat treatment.
6. Female patients who are pregnant or breast feeding, or without pregnancy test prior to Day 1.
7. History of significant lactose intolerance.
8. Clinically significant diarrhea (>3 liquid stools per day for >7 days) without definable cause within 6 months prior to Day 1, or a history of clinically relevant gastrointestinal disorders.
9. History of cataracts or known increased risk of cataract formation.
10. Severe renal impairment i.e., with a creatinine clearance <30 ml/min/1.73m^2
11. Concomitant active medical condition such as human immunodeficiency virus (HIV) or hepatitis B/C that would render patients unsuitable for study.
12. Previous treatment with miglustat.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-02-01; Primary Completion 2010-06-01 (Actual); Study Completion 2010-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Cox, Prof, Principal Investigator — University of Cambridge

REFERENCES:
- [Result] Cox TM, Amato D, Hollak CE, Luzy C, Silkey M, Giorgino R, Steiner RD; Miglustat Maintenance Study Group. Evaluation of miglustat as maintenance therapy after enzyme therapy in adults with stable type 1 Gaucher disease: a prospective, open-label non-inferiority study. Orphanet J Rare Dis. 2012 Dec 27;7:102. doi: 10.1186/1750-1172-7-102. PMID 23270487

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 16 centers in 10 countries (Australia, Brazil, Canada, Czech Republic, France, Netherlands , Spain, Taiwan, UK, and USA. The first patient, first visit was 21 February 2006 and the last patient, last visit was 22 June 2010.
Groups:
- Miglustat: Oral administration of miglustat 100 mg t.i.d. for a period of 2 years
Period: Overall Study
Arm/Group | Miglustat
Started | 42 (One patient was excluded from analysis as the baseline liver volume not available)
Completed | 34
Not Completed | 8
Not completed — withdrawal of subject's consent | 7
Not completed — administrative reason | 1

BASELINE CHARACTERISTICS:
Arm/Group | Miglustat
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (12.7)
Age, Customized [Number; unit: participants]
  Between 22 and 70 years | 42
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 22
Region of Enrollment [Number; unit: participants]
  Australia | 3
  Brazil | 1
  Canada | 5
  Czech Republic | 2
  France | 1
  Netherlands | 3
  Spain | 2
  Taiwan | 1
  United Kingdom | 6
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Liver Volume at Baseline and at End of Treatment
Description: Liver volume was assessed at baseline and end of treatment by magnetic resonance imaging. Imputation methods for patients with missing values at Month 24 were applied as follows: if a patient had at least 640 days of treatment with the study drug, the last observation that was not more than 2 days after the end of treatment was carried forward. If a patient had discontinued study drug before Day 640, the 'worst' within-patient value not more than 2 days after the end of treatment was used to impute the missing value.
Time Frame: Baseline and end of treatment (Month 24)
Population: One patient was excluded from analysis as the baseline liver volume not available
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Miglustat
Number analyzed (Participants) | 41
cm^3
  Baseline | 1774.6 (484.07)
  End of treatment | 1727.1 (381.73)

2. Primary Outcome: Mean Within-patient Percent Change From Baseline in Liver Volume
Description: as for outcome 1
Time Frame: End of treatment (Month 24)
Population: One patient was excluded from analysis as the baseline liver volume not available
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Miglustat
Number analyzed (Participants) | 41
Percentage change | -1.1 (13.75)

3. Secondary Outcome: Spleen Volume at Baseline and End of Treatment
Description: Spleen volume was assessed at baseline and end of treatment by magnetic resonance imaging.
  Imputation methods for patients with missing values at Month 24 were applied as follows: if a patient had at least 640 days of treatment with the study drug, the last observation that was not more than 2 days after the end of treatment was carried forward. If a patient had discontinued study drug before Day 640, the 'worst' within-patient value not more than 2 days after the end of treatment was used to impute the missing value.
Time Frame: Baseline and end of treatment (Month 24)
Population: The analysis was performed on those non-splenectomized patients who had a post-baseline assessment of spleen volume while on treatment with miglustat
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Miglustat
Number analyzed (Participants) | 22
cm^3
  Baseline | 509.8 (371.77)
  End of treatment | 611.9 (442.44)

4. Secondary Outcome: Mean Percent Change From Baseline in Spleen Volume
Description: as for outcome 3
Time Frame: End of treatment (Month 24)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Miglustat
Number analyzed (Participants) | 22
Percentage change | 21.1 (25.37)

ADVERSE EVENTS:
Time Frame: From study treatment start to the study treatment end date plus 2 days
Groups:
- Miglustat: Oral administration of miglustat 100 mg t.i.d. (median time exposure = 658 days)
Arm/Group | Miglustat
Serious Adverse Events (participants affected / at risk) | 5/42
Other Adverse Events (participants affected / at risk) | 40/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Miglustat (N=42)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
BLOOD URINE PRESENT (Investigations) | 1
CEREBELLAR SYNDROME (Nervous system disorders) | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CYST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 1
HYPERREFLEXIA (Nervous system disorders) | 1
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1
PNEUMONIA (Infections and infestations) | 1
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Miglustat (N=42)
DIARRHOEA (Gastrointestinal disorders) | 31
FLATULENCE (Gastrointestinal disorders) | 21
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 4
ABDOMINAL PAIN (Gastrointestinal disorders) | 4
NAUSEA (Gastrointestinal disorders) | 4
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3
TREMOR (Nervous system disorders) | 15
HEADACHE (Nervous system disorders) | 9
PARAESTHESIA (Nervous system disorders) | 9
DIZZINESS (Nervous system disorders) | 7
HYPOAESTHESIA (Nervous system disorders) | 5
CHITOTRIOSIDASE INCREASED (Investigations) | 6
WEIGHT DECREASED (Investigations) | 6
PLATELET COUNT DECREASED (Investigations) | 5
HAEMOGLOBIN DECREASED (Investigations) | 4
ANGIOTENSIN CONVERTING ENZYME INCREASED (Investigations) | 3
BLOOD FOLATE DECREASED (Investigations) | 3
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 4
BONE PAIN (Musculoskeletal and connective tissue disorders) | 3
NASOPHARYNGITIS (Infections and infestations) | 4
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4
FATIGUE (General disorders) | 8
DEPRESSION (Psychiatric disorders) | 3
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4
ANAEMIA (Blood and lymphatic system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less